CLINICAL TRIAL: NCT05197803
Title: Clinical Study of Released Unitron RIC (Receiver in Canal) and BTE (Behind the Ear) Hearing Aid Models
Brief Title: Clinical Study of Released Unitron RIC and BTE Hearing Aid Models
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Collaborators: Sonova Canada Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 515
Record Dates: First submitted 2021-12-16; First posted 2022-01-20 (Actual); Results first posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2023-11

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss | interventions — Hearing Aids

STUDY DESIGN:
Intervention Model Description: One similar intervention; 2 groups based on hearing aid model.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): The same group of participants undergo the same testing conditions. Each participant is fit with the BTE and the RIC hearing aids and then complete the speech intelligibility testing - Hearing in Noise Test (HINT) - aided and unaided during one-time visit.
  Interventions: Device: Hearing aid

INTERVENTIONS:
Device: Hearing aid — Participants will complete testing aided and unaided. The hearing aids have been fit to compensate for their hearing loss.

SUMMARY:
The present study will confirm the clinical benefit of 2 different released hearing aid models for speech understanding (in noise). Participants with mild to severe hearing impairment will be fit binaurally with Unitron hearing aids and will perform a standardized speech discrimination test in noise with and without hearing aids.

DETAILED DESCRIPTION:
Each participant will be asked to wear a set of BTE and RIC hearing aids and complete the Hearing in Noise Test (HINT) aided and unaided. The investigators will be assessing their speech intelligibility in noise for each condition during the same appointment to determine the SNR50 (the Signal-to-Noise ratio necessary for a participant to recognize the speech material correctly 50 percent of the time).

ELIGIBILITY:
Inclusion Criteria:

* Adults (18+ years) with hearing impairment (N2 - N6 hearing loss).
* Healthy outer ear.
* Symmetrical hearing loss.
* Ability to answer questions and repeat sentences.
* Informed consent as documented by signature.
* Willingness to wear different style of hearing aids.
* Willingness to wear a binaural fitting.
* Willingness to wear closed domes.
* Willingness to adhere to COVID protocols including correct mask use, completing screening for each visit

Exclusion Criteria:

* Contraindications to the medical device (MD) in this study (e.g. known hypersensitivity or allergy to the investigational product).
* Limited mobility/not able to come to scheduled visits.
* Inability to produce reliable hearing test result.
* Visible congenital or traumatic deformity of the outer ear.
* History of active drainage from the ear in the previous 90 days.
* Abnormal appearance of the eardrum and ear canal.
* Acute or chronic dizziness.
* Audiometric air-bone gap equal to or greater than 15 dB at 500 Hz, 1000 Hz, 2000 Hz, and 4000 Hz.
* Known psychological problems.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jinyu Qian, PhD, Principal Investigator — jinyu.qian@sonova.com
Locations (1):
- Unitron Hearing, Kitchener, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the existing participant local database. The first participant was enrolled on January 10, 2022 and the last participant was enrolled on January 28, 2022.
Pre-assignment Details: All 25 participants enrolled met the inclusion criteria established for this study.
Groups:
- Experimental: The same group of participants undergo one similar intervention. Each participant is fit with the BTE and the RIC hearing aids and then complete the speech intelligibility testing aided and unaided.
Period: Overall Study
Arm/Group | Experimental
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The same group of 25 participants undergo one similar intervention
Groups:
- Experimental: All participants are fit with the BTE and the RIC hearing aids and then complete speech intelligibility testing aided and unaided.
Arm/Group | Experimental
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.36 (11.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 25
Speech Intelligibility in Noise [Mean (Standard Deviation); unit: decibels (dB) Signal-to-Noise Ratio] — Sentences are presented through a speaker in front of the participant's head. Background noise is presented through other seven speakers arranged around the participant. The senteces are presented at varying levels (both louder and softer) than the fixed level of the noise. The SNR50 is the Signal-to-Noise Ratio at which te participant can repeat 50% of the words correctly. For example, an SNR50 of +3 means that the participant repeated 50% of the words back correctly when the sentences were presented at a level that was 3dB louder than the noise. Lower scores indicate better performance.
  decibels (dB) Signal-to-Noise Ratio | 1.7 (2.4)

OUTCOME MEASURES:

1. Primary Outcome: Speech Intelligibility Test in Noise
Description: Sentences are presented through a speaker in front of the participant's head. Background noise is presented through other seven speakers arranged around the participant. The senteces are presented at varying levels (both louder and softer) than the fixed level of the noise. The SNR50 is the Signal-to-Noise Ratio (SNR) expressed in decibels (dB) at which the participant can repeat 50% of the words correctly. For example, an SNR50 of +3 means that the participant repeated 50% of the words back correctly when the sentences were presented at a level that was 3dB louder than the noise. Lower scores indicate better performance.
Time Frame: 2 hours appointment
Population: The data for two participants had to be removed from the final analysis. In both cases, the speech intelligibiliy test could not be completed in one or more study conditions.
Measure: Mean (Standard Deviation); unit: decibel (dB) Signal-to-Noise Ratio
Arm/Group | Experimental
Number analyzed (Participants) | 23
decibel (dB) Signal-to-Noise Ratio
  dB SNR unaided condition | 0.83 (3.43)
  dB SNR aided condition (BTE) | -2.49 (1.93)
  dB SNR aided condition (RIC) | -2.74 (2.13)
Statistical Analysis 1: Comparison: Experimental; The study compared the results between the unaided condition vs. aided condition (BTE); Test type: Superiority; p = 0.0001, t-test, 1 sided; Mean Difference (Final Values) = 3.32
Statistical Analysis 2: Comparison: Experimental; The study compared the results between the unaided condition vs. aided condition (RIC); Test type: Superiority; p = 0.0001, t-test, 1 sided; Mean Difference (Final Values) = 3.57

ADVERSE EVENTS:
Time Frame: 1 day
Description: Hearing instruments do not generally cause mortality or serious adverse events. All participants underwent testing under the study conditions during one day appointment session. Therefore, all participants are combined for the Adverse Events reported.
Groups:
- Experimental: All participants performed the HINT test in a sound room setting and SNR50 scores were obtained under the three study conditions.
Arm/Group | Experimental
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-01-04): https://cdn.clinicaltrials.gov/large-docs/03/NCT05197803/Prot_SAP_ICF_000.pdf